CLINICAL TRIAL: NCT02380365
Title: QT-Prolongation in Lung Transplantation
Acronym: TX-QTC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2602-2015
Record Dates: First submitted 2015-03-02; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Disorder Related to Lung Transplantation
Keywords: lung transplantation; electrocardiography; macrolides; QTc interval; arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Outpatients on the Waiting List and after Lung Transplantation: Electrocardiography
  Interventions: Device: Electrocardiography

INTERVENTIONS:
Device: Electrocardiography — Duration of intervention per patient/subject:
  5 min, observation 6 months

SUMMARY:
Experimental intervention: electrocardiography. Control intervention: none

Duration of intervention per patient/subject:

5 min, observation 6 months

Key inclusion criteria:

* outpatients after lung transplantation (single, double or combined)
* outpatients on the wait list for lung transplantation

Key exclusion criteria:

• no informed consent

DETAILED DESCRIPTION:
Primary endpoint:

• prevalence of significant QTc-interval prolongation (500 msec or above) after lung transplantation

Key secondary endpoint(s):

* prevalence of any QTc-interval prolongation (>440 msec ) after lung transplantation
* prevalence of PQ prolongation (200 msec sec or above) after lung transplantation
* prevalence of QRS prolongation (120 msec or above) after lung transplantation
* prevalence of QTc-prolonging drugs in drug regimen before and after lung transplantation
* influence of long-term neo-macrolide (e.g. azithromycin) on QTc interval after lung transplantation
* intra-individual difference of QTc interval before and after lung transplantation
* incidence of any QTc-interval prolongation(>440 msec ) after lung transplantation
* incidence of any QTc-interval prolongation (>440 msec or increase by 50msec or above) after initiation of new QTc prolonging drugs (especially neo-macrolides)
* reversal of QTc-interval prolongation (440 msec or lower or decrease by 50msec or above) after stopping any QTc prolonging drug
* Assessment of safety:
* Incidence of new onset heart rhythm disorder during 6 months of follow-up

ELIGIBILITY:
Inclusion Criteria:

* outpatients after lung transplantation (single, double or combined)
* outpatients on the wait list for lung transplantation

Exclusion Criteria:

* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Follow-up Patients after lung transplantation
Sampling Method: Non-Probability Sample
Enrollment: 720 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
prevalence of significant QTc-interval prolongation (500 msec or above) after lung transplantation | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Jens Gottlieb, MD, Principal Investigator — Hannover MS, Dpt Respiratory Medicine
Locations (1):
- Department of Respiratory Medicine, Medizinische Hochschule Hannover, Hanover, Germany